CLINICAL TRIAL: NCT00359437
Title: Satavaptan in the Prevention of Ascites Recurrence: a Double-blind, Randomised, Parallel-group Comparison of Satavaptan at 5 to 10 mg Daily Versus Placebo With Concomitant Diuretics in Patients With Recurrent Ascites Due to Cirrhosis of the Liver.
Brief Title: Satavaptan in the Prevention of Ascites Recurrence in Patients With Ascites Due to Cirrhosis of the Liver
Acronym: SPARe-1
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EFC4493; EUDRACT: 2006-000132-27; LTS10036
Record Dates: First submitted 2006-08-01; First posted 2006-08-02 (Estimated); Last update posted 2016-05-24 (Estimated); Status verified 2016-04

CONDITIONS: Ascites; Liver Cirrhosis
MeSH Terms: conditions — Ascites; Liver Cirrhosis | interventions — satavaptan

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Satavaptan (Experimental)
  Interventions: Drug: Satavaptan
- Placebo (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Satavaptan — oral administration once daily
  Other Names: SR121463B
  Arms: Satavaptan
Drug: placebo — oral administration once daily
  Arms: Placebo

SUMMARY:
Primary To evaluate the efficacy of satavaptan on top of diuretic drugs in reducing the recurrence of ascites.

Secondary To evaluate the tolerability and safety of satavaptan on top of diuretic drugs over a 52-week treatment period in participants with cirrhosis of the liver and recurrent ascites.

The one-year double blind placebo controlled period is extended up to 2 years in a long term safety study (PASCCAL-2).

ELIGIBILITY:
Inclusion Criteria:

* Participants with cirrhosis of the liver.
* Participants with recurrent ascites having undergone both of the following:

  * therapeutic paracentesis for the removal of ascites in the previous 24 hours with the removal of > 4 litres of fluid.
  * at least one other therapeutic paracentesis in the previous 3 months.

Exclusion Criteria:

* Participants with an existing functional transjugular intrahepatic portosystemic shunt (TIPS) or other shunt.
* Known hepatocellular carcinoma.
* Participants with ascites of cardiac origin or due to peritoneal infection (e.g. tuberculosis) or peritoneal carcinoma.
* Participants previously exposed to satavaptan in the past 12 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 501 (Actual)
Dates: Start 2006-07; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Number and time of recurrences of therapeutic paracenteses | up to 12 weeks

SECONDARY OUTCOMES:
Time from randomisation to first recurrence of ascites | study period
Increase in ascites | over 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: ICD CSD, Study Director — Sanofi
Locations (24):
- Sanofi-Aventis Administrative Office, Malvern, Pennsylvania, United States
- Sanofi-Aventis Administrative Office, San Isidro, Argentina
- Sanofi-Aventis Administrative Office, Macquarie Park, Australia
- Sanofi-Aventis Administrative Office, Diegem, Belgium
- Sanofi-Aventis Administrative Office, Sarajevo, Bosnia and Herzegovina
- Sanofi-Aventis Administrative Office, Sofia, Bulgaria
- Sanofi-Aventis Administrative Office, Laval, Canada
- Sanofi-Aventis Administrative Office, Zagreb, Croatia
- Sanofi-Aventis Administrative Office, Prague, Czechia
- Sanofi-Aventis Administrative Office, Paris, France
- Sanofi-Aventis Administrative Office, Berlin, Germany
- Sanofi-Aventis Administrative Office, Budapest, Hungary
- Sanofi-Aventis Administrative Office, Netanya, Israel
- Sanofi-Aventis Administrative Office, Milan, Italy
- Sanofi-Aventis Administrative Office, Kuala Lumpur, Malaysia
- Sanofi-Aventis Administrative Office, Porto Salvo, Portugal
- Sanofi-Aventis Administrative Office, Bucharest, Romania
- Sanofi-Aventis Administrative Office, Belgrade, Serbia
- Sanofi-Aventis Administrative Office, Singapore, Singapore
- Sanofi-Aventis Administrative Office, Midrand, South Africa
- Sanofi-Aventis Administrative Office, Seoul, South Korea
- Sanofi-Aventis Administrative Office, Barcelona, Spain
- Sanofi-Aventis Administrative Office, Taipei, Taiwan
- Sanofi-Aventis Administrative Office, Guildford Surrey, United Kingdom

REFERENCES:
- [Derived] Wong F, Watson H, Gerbes A, Vilstrup H, Badalamenti S, Bernardi M, Gines P; Satavaptan Investigators Group. Satavaptan for the management of ascites in cirrhosis: efficacy and safety across the spectrum of ascites severity. Gut. 2012 Jan;61(1):108-16. doi: 10.1136/gutjnl-2011-300157. Epub 2011 Aug 11. PMID 21836029